CLINICAL TRIAL: NCT03510026
Title: Skeletonized Internal Thoracic Artery Harvesting: A Low Thermal Electrosurgical Device Provides Improved Endothelial Layer and Better Integrity of the Vessel Wall
Brief Title: Low Thermal Electrosurgical Device for Atraumatic Internal Thoracic Artery Harvesting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Alicja Zientara, Dr. med., Triemli Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2013-0017
Record Dates: First submitted 2018-04-04; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Preparation of Internal Thoracic Artery
Keywords: internal thoracic artery harvesting; arterial graft patency; electrosurgery; arterial graft preparation
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low thermal device preparation (Other): One participant acts simultaneously as a control and active comparator. One internal thoracic artery is prepared with the normal electrocautery device. The other internal thoracic artery is prepared with the new low thermal device. The participant does not know, which internal thoracic artery is defined to be prepared with the low thermal device.
  Interventions: Device: Low thermal device preparation

INTERVENTIONS:
Device: Low thermal device preparation — One participant acts simultaneously as a control and active comparator. One internal thoracic artery is prepared with the normal electrocautery device. The other internal thoracic artery is prepared with the new low thermal device. The participant does not know, which internal thoracic artery is defined to be prepared with the low thermal device.

SUMMARY:
Electrosurgery is fundamental to the precise, fast and bloodless preparation of internal thoracic artery grafts in cardiac surgery. The PEAK PlasmaBlade is a monopolar electrosurgical device that uses pulsed radiofrequency energy to generate a plasma-mediated discharge along an insulated electrode, creating a cutting edge while the blade stays near body temperature. The aim of this study is to compare the histological samples, cardiac computed-tomography of graft patency, and clinical outcomes of patients after off-pump coronary artery bypass grafting with preparation of the internal thoracic arteries by a conventional electrosurgical device and the PlasmaBlade.

DETAILED DESCRIPTION:
Electrosurgery is fundamental to the precise, fast and bloodless preparation of internal thoracic artery grafts in cardiac surgery. The fundamental performance of electrosurgical dissection is created by using a continuous radiofrequency energy waveform, which thermally ablates soft tissue, leaving a collateral damage zone of 100-400 µm. The basic mechanism of tissue ablation and dissection in electrosurgery involves Joule heating of the conductive tissue by electric current, that leads to vaporization and ionization of the water content in the tissue adjacent to the electrode, and ultimately to vapor expansion and tissue fragmentation. Tissue heated below the vaporization threshold remains in place, but can undergo thermal denaturation determined by the temperature levels and duration of the hyperthermia. Thus, to confine the collateral damage zone in tissue, both of these factors should be minimized.

In contrast to continuous radiofrequency energy, pulsed electric waveforms with burst durations ranging from 10 to 100 µsec applied via an insulated planar electrode with 12 µm wide exposed edge produces a plasma-mediated, precise dissection of tissues with a lower collateral damage zone ranging from 2 to 10 µm. The greatly reduced zone of thermal damage, compared to conventional electrosurgical devices, may provide faster healing and less scarring.

The PEAK PlasmaBlade (Medtronic Advanced Energy, Portsmouth, NH USA) (FDA 510(k), CE-No. 540861, Model Number PS200-040) is an electrosurgical device that uses pulsed radiofrequency energy to generate a plasma-mediated discharge along the exposed rim of an insulated blade, creating an effective, precise cutting edge while the blade stays near body temperature. Plasma is an electrically conductive cloud created when the energy contacts tissue. This conductive cloud or "plasma" allows the radiofrequency energy to cross at much lower overall power levels. This use of less energy via plasma results in lower operating temperatures and less thermal damage. This technology has been shown to effectively dissect ophthalmologic and cutaneous tissues as precisely as a scalpel with the hemostatic control of conventional electrosurgery in clinical and experimental settings.

Concentrating on bypass grafts, the thoracic internal arteries (ITAs) demonstrate our most valuable conduit for revascularization of the coronary arteries. Compared to pedicled arteries, skeletonized ITAs have demonstrated a tendency to better long term patency. Additionally, skeletonized conduits are useful in expanding the number of anastomoses per patient and reducing the incidence of sternal complications.

The use of a dissection device that provides precise preparation, including optimal bleeding control without overly damaging the surrounding tissue, might be an optimizing factor for the protection of these valuable bypass grafts. The aim of this study was to compare the histological assessment, cardiac computed-tomography and clinical outcomes of patients following off-pump coronary artery bypass grafting with preparation of the ITAs by conventional electrosurgery and the PlasmaBlade.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving elective coronary artery bypass grafting with both internal thoracic arteries
* signed consent

Exclusion Criteria:

* emergency procedures
* patients, who are already involved in other studies
* pregnant women or women of childbearing Age
* missing signed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08-08 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Endothelial damage | six months
  Histological examination of internal thoracic artery samples stained for endothelial damage.

SECONDARY OUTCOMES:
Vessel wall integrity | six months
  Histological examination of internal thoracic artery samples stained for vessel wall integrity.
Patency of internal thoracic arteries as bypass grafts | six months
  Computed tomography six months after bypass operation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zientara A, Komminoth P, Seifert B, Odavic D, Dzemali O, Haussler A, Genoni M. Skeletonized internal thoracic artery harvesting: a low thermal damage electrosurgical device provides improved endothelial layer and tendency to better integrity of the vessel wall compared to conventional electrosurgery. J Cardiothorac Surg. 2018 Oct 11;13(1):105. doi: 10.1186/s13019-018-0797-3. PMID 30305183